CLINICAL TRIAL: NCT04980534
Title: Evaluation of the Effectiveness of Therapy for Patients With Covid-19 Using Food Supplements Viusid + Asbrip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: COVID_KAZ_2021
Record Dates: First submitted 2021-07-26; First posted 2021-07-28 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2021-07

CONDITIONS: Covid19; COVID-19 Pneumonia; COVID-19 Respiratory Infection; Viral Infection; Respiratory Tract Infections; Infection, Coronavirus; SARS-CoV2 Infection
Keywords: covid-19; supportive care; Immuno-modulator; antiviral; symptoms relieve
MeSH Terms: conditions — COVID-19; Virus Diseases; Respiratory Tract Infections; Coronavirus Infections | interventions — Viusid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Viusid Plus Asbrip Adjuvant (Experimental): 25 Patients who received standard therapy Remdesivir IV 200 mg for the first day and then 100 mg daily for the next 4 days AND Viusid (sachets with powder for dilution, oral administration) 1 sachet bid and Asbrip (liquid form, oral administration) 10 ml bid for the total duration of hospitalization. Time Frame: 21 days.
  Interventions: Dietary Supplement: Viusid and Asbrip; Drug: COVID-19 Standard Therapy
- Viusid Plus Asbrip Monotherapy (Experimental): 25 Patients who did not receive standard antiviral therapy with the inclusion of food supplements Viusid (4.5 gr every 12 hours, oral administration) and Asbrip (10 mL every 12 hours, oral administration). Time Frame: 21 days.
  Interventions: Dietary Supplement: Viusid and Asbrip
- Control (Active Comparator): 30 patients who received standard therapy (Remdesivir IV 200 mg for the first day and then 100 mg daily for the next 4 days), without the inclusion of food supplements Viusid and Asbrip.
  Interventions: Drug: COVID-19 Standard Therapy

INTERVENTIONS:
Dietary Supplement: Viusid and Asbrip — Patients will be assigned to receive daily oral doses of 4.5gr of Viusid and 10 ml of Asbrip every 8 hours and standard care.
  Arms: Viusid Plus Asbrip Adjuvant; Viusid Plus Asbrip Monotherapy
Drug: COVID-19 Standard Therapy — Patients will be assigned to receive the standard therapy for COVID-19 disease: Antibiotic, Antivirals, Analgaesic, Anti-inflammatory drugs.
  Arms: Control; Viusid Plus Asbrip Adjuvant

SUMMARY:
This is a two-arm, randomized, open label, monocenter, controlled study to evaluate the safety and efficacy of Viusid plus Asbrip in patients with mild and moderate symptoms of respiratory illness caused by Coronavirus 2019 infection.

DETAILED DESCRIPTION:
This is a two-arm, randomized, open label, monocenter, controlled study to evaluate the safety and efficacy of Viusid plus Asbrip in patients with mild and moderate symptoms of respiratory illness caused by Coronavirus 2019 infection.

A total of 80 subjects will be randomized 2:1 in this study. 50 patients will be assigned to receive daily oral doses of 4,5 g of Viusid every 12 hours and 10 ml of Asbrip every 12 hours and standard care with antivirals or not. Other 30 patients will be assigned to receive only standard care.

Treatment duration: 21 days

Objective of the study: to increase the effectiveness of therapy for patients with Covid-19 using food supplements Viusid and Asbrip.

Research objectives:

1. To assess the clinical symptoms of Covid-19 in patients on the background of combination therapy with the inclusion of food supplements Viusid + Asbrip.
2. To investigate the dynamics of indicators of laboratory diagnostics against the background of complex therapy with the inclusion of food additives Viusid + Asbrip in the complex treatment of Covid -19.
3. To study the dynamics of indicators of instrumental methods of treatment.
4. To develop an algorithm for the management of patients with coronavirus infection in order to increase the effectiveness of therapy and rehabilitation of patients with this pathology.

ELIGIBILITY:
The eligibility criteria for inclusion in the study were as follows:

* Male and female hospitalized patients who have signed an informed consent.
* Aged between 18-85 years old.
* RT-PCR confirmed COVID-19.
* Fever (over 37.2 Celsius degrees).
* CT scan percentage area of lung involvement with ground-glass opacities < 50 %.
* Respiratory rate < 20-30 /min
* SpO2 ≥ 95%.

The exclusion criteria were as follows:

* Oxygen support (ventilation and non-invasive)
* Uncompensated or exacerbated concomitant diseases or conditions that may complicate or make the patient's participation in the study impossible, or make it difficult to explain clinical findings.
* Any known intolerability to any of the study regimens' components.
* Patient's family or official relations with a member of staff of the clinical site.
* Patient's failure to assess his/her physical and/or emotional condition.
* Patient's failure to comply with the study requirements.
* Patient's refusal to participate in the study.
* Pregnancy or breastfeeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Mean duration of hospitalization. | 21 days
  Media of time in days to discharge in each group. Discharge is considered once the patient complete the following conditions:
  * Normal body temperature for 2 days (36.1 - 37.2 degrees Celsius will be considered as normal body temperature).
  * Normal appetite for 4 days.
  * Normal Complete Blood Count (CBC): Following values will be considered as normal values in CBC:
  Red blood cell count: Male: 4.35-5.65 million cells/mcL; Female: 3.92-5.13 million cells/mcL. Hemoglobin: Male: 13.2-16.6 grams/dL; Female: 11.6-15 grams/dL. Hematocrit: Male: 38.3-48.6 percent; Female: 35.5-44.9 percent. White blood cell count: 3,400 to 9,600 cells/mcL. Platelet count: Male: 135-317 billion/L; Female: 157-371 billion/L.
  * No requirement in oxygen support.
  * Decrease in or normal CRP: 0.8-1.0 mg/dL (or 8-10 mg/L) or lower will be considered as normal values.
  * Any decrease in IL-6 level lower than doubled normal value: between 0 and 43.5 pg/ml will be considered as normal values.

SECONDARY OUTCOMES:
Mean levels of IL-6 concentration | 21 days
  Mean of IL-6 concentration measured by blood biochemical analysis at day 0, 5, 10, 15 and 21. IL-6 level lower than doubled normal value: between 0 and 43.5 pg/ml will be considered as normal values.
  Levels of IL-6 will be determined centrally at OLYMP diagnostics lab (https://www.kdlolymp.kz/).
Peripheral blood c-reactive protein concentration | 21 days
  Peripheral blood c-reactive protein concentration measured by blood biochemical analysis at day 0, 5, 10, 15 and 21.
  - 0.8-1.0 mg/dL (or 8-10 mg/L) or lower will be considered as normal values.
  Levels of CRP will be determined centrally at OLYMP diagnostics lab (https://www.kdlolymp.kz/).
Mean levels of D-Dimer concentration | 21 days
  Mean of D-dimer measured by blood biochemical analysis at day 0, 5, 10, 15 and 21. D-Dimer level under 250 ng/mL, or under 0.4 μ/mL will be considered as normal value.
  Levels of D-Dimer will be determined centrally at OLYMP diagnostics lab (https://www.kdlolymp.kz/).
Mean levels of Ferritin concentration | 21 days
  Mean of D-dimer measured by blood biochemical analysis at day 0, 5, 10, 15 and 21. In adult Males between 12 to 300 ng/mL; in adult Females between 12 to 150 ng/mL will be considered as normal values.
  Levels of Ferritin will be determined centrally at OLYMP diagnostics lab (https://www.kdlolymp.kz/).

CONTACTS AND LOCATIONS:
Locations (3):
- Kazakhstan (3):
  - City center for infectious diseases, Astana, Astana
  - City children hospital №1, Astana, Astana
  - JSC "Astana Medical University, Astana

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621
- [Result] Gomez EV, Perez YM, Sanchez HV, Forment GR, Soler EA, Bertot LC, Garcia AY, del Rosario Abreu Vazquez M, Fabian LG. Antioxidant and immunomodulatory effects of Viusid in patients with chronic hepatitis C. World J Gastroenterol. 2010 Jun 7;16(21):2638-47. doi: 10.3748/wjg.v16.i21.2638. PMID 20518086
- [Result] Vilar Gomez E, Rodriguez De Miranda A, Gra Oramas B, Arus Soler E, Llanio Navarro R, Calzadilla Bertot L, Yasells Garcia A, Del Rosario Abreu Vazquez M. Clinical trial: a nutritional supplement Viusid, in combination with diet and exercise, in patients with nonalcoholic fatty liver disease. Aliment Pharmacol Ther. 2009 Nov 15;30(10):999-1009. doi: 10.1111/j.1365-2036.2009.04122.x. Epub 2009 Aug 18. PMID 19691668
- See also: Related Info — https://www.researchgate.net/publication/340522164_Nueva_alternativa_para_el_tratamiento_para_Covid_19_en_Ecuador
- See also: Related Info — https://clinicaltrials.gov/ct2/show/NCT04407182
- See also: Related Info — https://www.hilarispublisher.com/open-access/effectiveness-of-viusid-and-asbrip-in-hospitalized-patients-infected-by-sarscov2-and-mildtomoderate-respiratory-illness-.pdf